CLINICAL TRIAL: NCT04916366
Title: Efficacy of Kinesio Taping in Musculoskeletal Neck Pain in Short and Medium Term. A Randomized Control Double Blinded Clinical Trial
Brief Title: Efficacy of Kinesio Taping in Musculoskeletal Neck Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 18/133-E_TFG
Record Dates: First submitted 2021-06-02; First posted 2021-06-07 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Musculoskeletal Neck Pain
Keywords: Musculoskeletal Neck Pain; Kinesio Taping

STUDY DESIGN:
Intervention Model Description: A double-blind controlled clinical trial.
Who Masked: Participant, Care Provider, Investigator
Masking Description: An investigator will carried out the measurement of the baseline variables. An expertise physiotherapy with experience in kinesio taping application, will performed the intervention with Kinesio taping in neck.
  All patients will be told that they are going to undergo a kinesio taping treatment, except for the control group, which will be given the option of being included in the experimental group once the follow-up process is over.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Kinesio taping (Experimental): In this arm, patients will be treated with blue Kinesio taping in a muscle relaxation position during 4 days.
  Interventions: Other: Kinesio taping
- Placebo (Placebo Comparator): In this arm, patients will be treated with conventional bandage in a muscle relaxation position during 4 days.
  Interventions: Other: Conventional bandage
- Control (No Intervention): In this arm, patients will be not treated but the outcomes will be measure after 4 days.

INTERVENTIONS:
Other: Kinesio taping — Kinesio taping in a bandage to treat musculoskeletal pain.
  Arms: Kinesio taping
Other: Conventional bandage — It will be used a conventional bandage applicated in the same neck region than kinesio taping intervention.
  Arms: Placebo

SUMMARY:
The aim of this study is to compare efficacy of Kinesio taping against a conventional tape in a patient with cervical musculoskeletal pain. For this, a double-blind controlled clinical trial be carried out in patients with musculoskeletal neck pain.

DETAILED DESCRIPTION:
During the months of May to July 2021, a research assistant will contact potential participants who will be invited to participate in this study. Once they agree to participate, it will schedule for a face-to-face consultation at the university, where the main researcher will inform the study participants. Once the information sheet and informed consent will be a sign, an investigator will carry out the measurements of the variables for initial data collection in the first session. In another room, an expertise physiotherapist with experience in applying Kinesio taping will perform interventions on patients on the same day as the initial evaluation. It this way, the investigator that will assess outcomes will be blind to the treatment that each patient will receive.

At the second consultation, 4 days after the first, the same physiotherapist who applied the bandage will remove it from the patients who received it and any remains of the bandage on the skin were cleaned. For patients in the control group (nothing apply), it will be the same protocol to alter, not the double-blind. The principal investigator will perform the evaluations and data collection without knowing the intervention the patient will receive.

In a third consultation, as a follow-up (30 days after the second consultation), the collection of the same measurements and clinical variables from the patients who completed the process will repeat by the same investigator that did the outcomes' assessment.

ELIGIBILITY:
Inclusion Criteria:

* Presence of myofascial pain syndrome (MPS) and myofascial trigger point (MTP) in the upper trapezius muscle, according to the diagnostic criteria proposed by the American Academy of Pain Medicine(2) and the scientific community (3) a) tender point on palpation, with or without referred pain b) patient recognizes pain during tender point palpation c) at least three of the following: muscle stiffness or muscle spasm, limited range of motion in an associated joint, increase of pain with stress, palpation of tight band and / or nodule, associated with a tender point
* understand written Spanish.

Exclusion Criteria:

* Neck pain of traumatic origin, due to recent surgery or causing radiculopathy
* Have been diagnosed with chronic pathology, as well as neoplastic or suspicion of it
* Have received some type of pharmacological or non-pharmacological analgesic treatment in the last 30 days.
* Pregnant or menstrual women

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Baseline Pain intensity | Baseline
  assessed by numerical rating scale (NRS) (5). Self-evaluation system of a scale with scores from "0" to "10", where "0" = absence of pain and "10" = maximum pain tolerable by the patient. A value lower than 4 means "mild pain, a value between 4-6 moderate pain, and values of 6-10 implies the presence of intense pain
Post-treatment Pain intensity | 4 days after treatment
  assessed by numerical rating scale (NRS) (5). Self-evaluation system of a scale with scores from "0" to "10", where "0" = absence of pain and "10" = maximum pain tolerable by the patient. A value lower than 4 means "mild pain, a value between 4-6 moderate pain, and values of 6-10 implies the presence of intense pain
Follow-up Pain intensity | 30 days after treatment
  assessed by numerical rating scale (NRS) (5). Self-evaluation system of a scale with scores from "0" to "10", where "0" = absence of pain and "10" = maximum pain tolerable by the patient. A value lower than 4 means "mild pain, a value between 4-6 moderate pain, and values of 6-10 implies the presence of intense pain
Baseline Health-related quality of life | Baseline
  assessed using the Short Form-36 (SF-36) questionnaire (6). This is a 36-item self-evaluating instrument where the perception of physical and emotional health is assessed in the 4 weeks before taking the questionnaire. The score ranges from "0" to "100", where a higher score implies a higher grade in health-related quality of life. This questionnaire has been shown to have adequate psychometric quality
Post-treatment Health-related quality of life | 4 days after treatment
  assessed using the SF-36 questionnaire (6). This is a 36-item self-evaluating instrument where the perception of physical and emotional health is assessed in the 4 weeks before taking the questionnaire. The score ranges from "0" to "100", where a higher score implies a higher grade in health-related quality of life. This questionnaire has been shown to have adequate psychometric quality
Follow-up Health-related quality of life | 30 days after treatment
  assessed using the SF-36 questionnaire (6). This is a 36-item self-evaluating instrument where the perception of physical and emotional health is assessed in the 4 weeks before taking the questionnaire. The score ranges from "0" to "100", where a higher score implies a higher grade in health-related quality of life. This questionnaire has been shown to have adequate psychometric quality
Baseline Impact of neck pain on daily life | Baseline
  assessed using the Neck Pain Questionnaire (NPQ)(7). It is made up of 9 items, which can be answered using a 5-response Likert scale. The result is represented in percentage values, where higher percentage means/shows more significant and negative impact on the patient's daily actions. The questionnaire has been validated in the Spanish language and population, showing adequate validity and reliability
Post-treatment Impact of neck pain on daily life | 4 days after treatment
  assessed using the Neck Pain Questionnaire (NPQ)(7). It is made up of 9 items, which can be answered using a 5-response Likert scale. The result is represented in percentage values, where higher percentage means/shows more significant and negative impact on the patient's daily actions. The questionnaire has been validated in the Spanish language and population, showing adequate validity and reliability
Follow-up Impact of neck pain on daily life | 30 days after treatment
  assessed using the Neck Pain Questionnaire (NPQ)(7). It is made up of 9 items, which can be answered using a 5-response Likert scale. The result is represented in percentage values, where higher percentage means/shows more significant and negative impact on the patient's daily actions. The questionnaire has been validated in the Spanish language and population, showing adequate validity and reliability
Baseline Pressure pain threshold (PPT) | Baseline
  Assessed by pressure algometry. Assesses the minimum pressure necessary to trigger an uncomfortable sensation associated with pain(8). This method is valid and reliable to measure the sensitivity of an MTP if three consecutive measurements are made and allowing a rest time between 30 seconds to 1 minute between measurements.Algometer has demonstrated an inter-examiner reliability range of 0.91(95% Interval coefficient CI)), showing adequate reliability for research if performed by inexperienced evaluators (9). The PPT is expressed in kPa (kilopascal), for an accurate evaluation, the force to be applied with algometer must be perpendicular to the point to be measured, without the skin sliding over the subcutaneous tissue. And a constant force must be applied, currently the application of a constant force with an acceleration of 5kPa is advocated (8). The PPT was measured in the MTP 2 of the upper trapezius, taking three measurements and taking the arithmetic mean of the three.
Post-treatment Pressure pain threshold (PPT) | 4 days after treatment
  Assessed by pressure algometry. Assesses the minimum pressure necessary to trigger an uncomfortable sensation associated with pain(8). This method is valid and reliable to measure the sensitivity of a MTP if three consecutive measurements are made and allowing a rest time between 30 seconds to 1 minute between measurements. Algometer has demonstrated an inter-examiner reliability range of 0.91 (95% CI, 0.82-0.97), showing adequate reliability for research if performed by inexperienced evaluators (9). The PPT is expressed in kPa (1kg / cm2 = 98.0665 kPa), for an accurate evaluation, the force to be applied with the algometer must be perpendicular to the point to be measured, without the skin sliding over the subcutaneous tissue. and a constant force must be applied, currently the application of a constant force with an acceleration of 5kPa is advocated (8). The PPT was measured in the MTP 2 of the upper trapezius, taking three measurements and taking the arithmetic mean of the three.
Follow-up Pressure pain threshold (PPT) | 30 days after treatment
  Assessed by pressure algometry. Assesses the minimum pressure necessary to trigger an uncomfortable sensation associated with pain(8). This method is valid and reliable to measure the sensitivity of a MTP if three consecutive measurements are made and allowing a rest time between 30 seconds to 1 minute between measurements. Algometer has demonstrated an inter-examiner reliability range of 0.91 (95% CI, 0.82-0.97), showing adequate reliability for research if performed by inexperienced evaluators (9). The PPT is expressed in kPa (1kg / cm2 = 98.0665 kPa), for an accurate evaluation, the force to be applied with the algometer must be perpendicular to the point to be measured, without the skin sliding over the subcutaneous tissue. and a constant force must be applied, currently the application of a constant force with an acceleration of 5kPa is advocated (8). The PPT was measured in the MTP 2 of the upper trapezius, taking three measurements and taking the arithmetic mean of the three.
Suggestibility | Baseline
  measured by the Inventor of Suggestibility questionnaire (IS) (10). It is made up of 22 items and 4 subconstructs: fantasizing, concentration, emotional involvement and influencing. It consists of 22 items with five-point Likert-type scalar response options ("0" = "almost never"; to "4" = "almost always"), where patients must respond about the frequency with which certain reactions appear in their daily life, with a high score being an indicator of greater suggestibility

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nurse, Physiotherapy and Podiatry. University Complutense of Madrid, Madrid, Spain

DOCUMENTS (2):
  • Study Protocol (2021-06-01): https://cdn.clinicaltrials.gov/large-docs/66/NCT04916366/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-01): https://cdn.clinicaltrials.gov/large-docs/66/NCT04916366/SAP_001.pdf